CLINICAL TRIAL: NCT06095882
Title: Randomized Controlled, Open Clinical Study on Efficacy and Safety of Acupuncture for Bladder Function Recovery After Radical Cervical Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202309-002
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Experimental)
  Interventions: Other: acupuncture
- observe (No Intervention)

INTERVENTIONS:
Other: acupuncture — Study group: Acupuncture treatment was performed from day 3 to day 14 after surgery. Points include: Zhongwan, Tianshu, Watercourse, Taichong, Sanyinjiao, Zusanli, Yin Lingquan.
  Control group: No intervention, the urinary tube was removed until the 14th day after surgery. Patients with urinary retention may receive further acupuncture treatment.
  Arms: acupuncture

SUMMARY:
Urinary retention is one of the most common complications of radical hysterectomy in patients with cervical cancer, with an incidence of 26-53% depending on the diagnostic criteria.

The most common method to prevent urinary retention after radical hysterectomy is continuous catheterization, but up to 14.5% of patients need continuous catheterization for more than 4 weeks, because catheterization is an invasive procedure, increasing the risk of urinary tract infection, and long-term postoperative retention of urinary catheter caused by edema of the vesicourethral sphincter and urethral glands. Obstruction of bladder outlet caused by increased urethral outflow resistance may also lead to postoperative urinary retention, thus forming a vicious cycle and aggravating urinary retention.

In our previous retrospective analysis, it was confirmed that acupuncture and moxibustion were effective in restoring bladder function after radical hysterectomy. Compared with the control group, the incidence of urinary retention in patients receiving acupuncture and moxibustion was reduced from 44.17% to 24.17%, and no serious adverse reactions occurred, and the patients had good tolerance. We plan to conduct further randomized controlled studies to confirm this.

DETAILED DESCRIPTION:
1. Basis for project establishment Cervical cancer is a deadly gynecological malignancy, with about 98,900 new cases and 30,500 deaths every year in China, and the age of onset is decreasing[1]. According to the 2022 NCCN guidelines, radical hysterectomy combined with pelvic lymphadenectomy is the standard surgical protocol for early cervical cancer, however, 30-85% of patients experience bladder dysfunction after radical hysterectomy, with negative effects on postoperative recovery and the patient's quality of life [2-4].

   Urinary retention is one of the most common complications of radical hysterectomy, with an incidence of 26-53% according to different diagnostic criteria [5-7], mainly due to bladder paralysis or dysfunction caused by amputation or injury of the bladder autonomic nerve, extensive excision of the sacral ligament, the major ligament, and the vagina [8-10]. In recent years, nerve sparing radical hysterectomy has received widespread attention, but due to the complex anatomy of the pelvic nerve, the difficulty of the operation, and more importantly, the incomplete resection of the tumor, this surgery has not been widely used in clinical practices[11]. Currently, the most commonly used method to prevent urinary retention after radical hysterectomy is continuous catheterization, but up to 14.5% of patients require continuous catheterization for more than 4 weeks, due to the invasive procedure, increasing the risk of urinary tract infection[12], and long-term postoperative indwelling of urinary tubes caused by vesicourethral sphincter and urethral gland edema. Obstruction of bladder outlet caused by increased urethral outflow resistance may also lead to postoperative urinary retention. This creates a vicious cycle that exacerbates urinary retention [13]. Therefore, the use of effective treatment means to strengthen the contraction ability of the detrusor muscle of the bladder and reduce spasm of the external urethral sphincter can help improve the bladder function impairment caused by surgery, restore the bladder urination function, reduce the pain of resetting the urinary tube and the probability of urinary system infection, and improve the quality of life of patients. For this reason, scholars have conducted some studies. Such as sacral neuromodulation [14,15] and drug therapy [16,17], however, have not achieved a very significant therapeutic effect. Therefore, it is necessary for us to further explore a better treatment to solve this clinical challenge.

   Acupuncture and moxibustion is an ancient treatment method originated in ancient China, which can be used to treat postoperative urinary retention from thousands of years of literature records and clinical practice. Previous studies have also confirmed its partial effect on urinary retention, [18-20], increasing the success rate of urinary tube removal, reducing the length of hospital stay, and alleviating patients' pain. In traditional Chinese medicine, urine retention after surgery is classified into the category of "retention of urine". The disease is located in the bladder, which is closely related to lung, spleen, kidney and three jiao. It is believed that the main mechanism of its occurrence is the injury of Chongren and other veins and the deficiency of qi and blood. Kidney deficiency leads to gasified disorganization and unfavorable bladder opening and closing. Spleen deficiency and dereliction of duty, water is not wet, eventually resulting in poor urine, urine retention.

   Through the previous study of modern acupuncture and moxibustion literature, we found that the common acupoints for preventing and treating urinary retention were mainly concentrated in the lower extremities, lower abdomen and lumbsacral area [21,22], such as Ciliao, Yinlingquan and Sanyinjiao, and the curative effect of Yinlingquan was superior to Sanyinjiao [23]. In our previous retrospective analysis, it was also confirmed that acupuncture was effective in restoring bladder function after radical hysterectomy. Compared with the control group, the incidence of urinary retention in patients receiving acupuncture was reduced from 44.17% to 24.17%, and no serious adverse reactions occurred, and the patient tolerance was good. In order to objectively observe the clinical therapeutic effect of acupuncture on the recovery of bladder function in patients after radical hysterectomy, we plan to further carry out randomized controlled studies to confirm, and analyze the characteristics and spatial distribution of tenderness sensitization, explore the correlation law of acupoint-zang-organ/body, and evaluate the specific connection difference between different acupoints and internal organs, so as to provide objective basis for clinical selection of acupoints.
2. Test purpose 2.1 Main research objectives: To evaluate the efficacy and safety of acupuncture for bladder function recovery after radical cervical cancer surgery by comparing the residual urine volume after catheter removal 14 days after surgery.

2.2 Secondary research purposes and exploratory research purposes:

1. To explore the characteristics and spatial distribution of acupoint tenderness sensitization of patients after radical cervical cancer surgery;
2. Explore the relevant laws of acupoint-zang-fu/body;
3. To explore the correlation between the occurrence of urinary retention and related clinicopathological features;
4. To explore the influence of acupuncture treatment on the prognosis of patients. 3. Pilot plan 3.1 Experimental design The objective of this study was to evaluate the residual urine volume of catheter removal 14 days after radical hysterectomy in patients with cervical cancer, and to evaluate the efficacy and safety of acupuncture for bladder function recovery after radical hysterectomy for cervical cancer.

A total of 180 patients with preoperative cervical lesions ≤4cm were randomly assigned to the observation group and acupuncture treatment group according to 1:1. The patients in the study group received acupuncture treatment from the 3rd day after surgery to the 14th day after surgery. The acupuncture points included Zhongwan, Tianshu, Shuitshui, Taichong, Sanyinjiao, Zusanli and Yin Lingquan. The control group had no intervention measures, and the urinary tube was removed on the 14th day after surgery. The control group patients with urinary retention could receive further acupuncture treatment.

The study was divided into screening period, treatment period and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1) The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with the follow-up; (2) Female, ≥18 years of age (calculated on the date of signing the informed consent); (3) Pathological diagnosis of cervical cancer, including squamous cell carcinoma, adenocarcinoma and adenosquamous cell carcinoma, preoperative cervical lesions ≤4cm; (4) No history of urinary system infection and urinary retention; (5) Undergoing radical abdominal hysterectomy; (6) On the third day after surgery, vital signs were stable, no discomfort symptoms (such as abnormal abdominal distension, nausea, vomiting, abdominal pain, chest tightness, etc.) of CTCAE 5.0 standard 2 or above, and no abnormal increase in body temperature (≥38.5°C); (7) The function of vital organs meets the following requirements: Absolute neutrophil count ≥1.5×109/L; Platelet ≥100×109/L; Hemoglobin ≥80g/L; Serum albumin ≥2.5g/dL; Bilirubin ≤1.5 ULN; ALT and AST≤3 times ULN; Serum creatinine ≤1.5 ULN; INR≤1.5 or prothrombin time ≤ULN+4 seconds.

Exclusion Criteria:

1. Suffering from diseases that may affect bladder function, such as uterine prolapse, vaginal wall bulge, lower urinary tract obstruction, bladder tumor, urethral injury, urinary tract stones, urinary tract infection, spinal cord injury, and sequelae of cardiovascular and cerebrovascular diseases;
2. Poor compliance and failure to strictly carry out full treatment;
3. Use of neostigmine and other drugs that affect bladder function;
4. Patients with serious diseases of important organs and mental diseases;
5. There were random postoperative discomfort symptoms with the severity reaching CTCAE 5.0 level 2 or above;
6. There is an active infection or prerandom unexplained fever ≥38.5°C;
7. Patients with clinical symptoms or diseases of heart that are not well controlled, such as: NYHA2 or above heart failure, unstable angina pectoris, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. diabetic patients;
9. In the judgment of the investigator, the subjects have other factors that may lead to the forced termination of the study, such as other serious diseases (including mental illness) requiring combined treatment, serious abnormalities in laboratory tests, and family or social factors that may affect the safety of the subjects or the collection of data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of urinary retention | 1year
  The urinary tube was removed 14 days after operation and the residual urine volume was measured